CLINICAL TRIAL: NCT03152812
Title: Functional Outcome of Free Muscle Flaps Versus Free Skin Flaps for Post-traumatic Foot Plantar Surface Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: alhussein Ahmed Mahmoud El-Dahshan (Other)
Responsible Party: Sponsor-Investigator, alhussein Ahmed Mahmoud El-Dahshan, Principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: salmaalhussein
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Best Tissue Constituent for Plantar Surface

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- free skin flaps
  Interventions: Procedure: plantar surface reconstruction by free flaps
- free muscle flaps
  Interventions: Procedure: plantar surface reconstruction by free flaps

INTERVENTIONS:
Procedure: plantar surface reconstruction by free flaps — use of free skin or free muscle flaps for reconstruction of plantar surface

SUMMARY:
the investigators are trying to detect what is the best tissue constituent suitable for reconstruction of large post traumatic sof tissue defects of foot plantar surface

ELIGIBILITY:
Inclusion Criteria:

1. Posttraumatic large soft tissue defects of plantar surface requiring free tissue transfer for coverage
2. At any age

Exclusion Criteria:

1-defects that can be managed by local flaps 2-Non traumatic soft tissue defects

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: any individual having post traumatic soft tissue defect of plantar surface requiring free flap reconstruction regardless to age
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Time to mobilize | 2 years
Requirement of specialized Footwear | 2 years

SECONDARY OUTCOMES:
flap ulceration | 2 years
Shear forces across the flap | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Amr El-Said Ali Ibrahim, MD, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No